CLINICAL TRIAL: NCT00143130
Title: Pregabalin in Partial Seizures (PREPS) Extension Study: An 18-month Follow-on Open-label, International, Multicenter Add-on Therapy Trial
Brief Title: Pregabalin In Partial Seizures Extension Study
Acronym: PREPS EXT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A0081015
Record Dates: First submitted 2005-08-31; First posted 2005-09-02 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2015-03

CONDITIONS: Seizures
Keywords: phase 4, open label, seizures, epilepsy, add-on therapy, pregabalin, lyrica
MeSH Terms: conditions — Seizures; Epilepsy | interventions — Pregabalin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: Pregabalin

INTERVENTIONS:
Drug: Pregabalin — Pregabalin

SUMMARY:
To evaluate long-term efficacy and safety of pregabalin (150 to 600mg/day) as adjunctive treatment in patients with partial seizures.

ELIGIBILITY:
Inclusion Criteria:

* met the inclusion/exclusion criteria for A0081005
* have completed the 21-week study and have shown a significant clinical response and wish to continue treatment

Exclusion Criteria:

* Having a treatable cause of seizure.
* Having a progressive neurological or systemic disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 2005-04; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Reduction in seizure frequency. | 18 months

SECONDARY OUTCOMES:
Seizure-free patients during each 3-month period | 18 Months
Responder Rate 50% during each 3-month period (proportion of patients with 50% or greater reduction of seizures). | 18 Months
Responder rate 75% during each 3-month period (proportion of patients with 75% or greater reduction of seizures). | 18 Months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (41):
- Belgium (8):
  - Pfizer Investigational Site, Bruges
  - Pfizer Investigational Site, Brussels
  - Pfizer Investigational Site, Duffel
  - Pfizer Investigational Site, Ghent
  - Pfizer Investigational Site, Leuven
  - Pfizer Investigational Site, Liège
  - Pfizer Investigational Site, Tielt
  - Pfizer Investigational Site, Yvoir
- Finland (3):
  - Pfizer Investigational Site, Helsinki
  - Pfizer Investigational Site, Kuopio
  - Pfizer Investigational Site, Tampere
- France (16):
  - Pfizer Investigational Site, Paris, Cedex 14
  - Pfizer Investigational Site, Lille, Cedex
  - Pfizer Investigational Site, Lyon, Cedex
  - Pfizer Investigational Site, Marsille, Cedex
  - Pfizer Investigational Site, Rennes, Cedex
  - Pfizer Investigational Site, Bayonne
  - Pfizer Investigational Site, Bordeaux
  - Pfizer Investigational Site, Grenoble
  - Pfizer Investigational Site, Marseille 13
  - Pfizer Investigational Site, Montpellier
  - Pfizer Investigational Site, Nancy
  - Pfizer Investigational Site, Nice
  - Pfizer Investigational Site, Paris
  - Pfizer Investigational Site, Strasbourg
  - Pfizer Investigational Site, Toulouse
  - Pfizer Investigational Site, Tours
- Poland (5):
  - Pfizer Investigational Site, Katowice
  - Pfizer Investigational Site, Krakow
  - Pfizer Investigational Site, Lublin
  - Pfizer Investigational Site, Warsaw
  - Pfizer Investigational Site, Wroclaw
- Portugal (7):
  - Pfizer Investigational Site, Braga
  - Pfizer Investigational Site, Coimbra
  - Pfizer Investigational Site, Funchal
  - Pfizer Investigational Site, Lisbon
  - Pfizer Investigational Site, Matosinhos Municipality
  - Pfizer Investigational Site, Ponta Delgada
  - Pfizer Investigational Site, Porto
- Switzerland (2):
  - Pfizer Investigational Site, Lausanne
  - Pfizer Investigational Site, Zurich

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081015&StudyName=Pregabalin%20In%20Partial%20Seizures%20Extension%20Study